CLINICAL TRIAL: NCT03268135
Title: Study of the Transcriptomic Alterations in Heart Failure and Aortic Stenosis
Brief Title: Heart Failure and Aortic Stenosis Transcriptome
Acronym: RNA-HF-AS
Status: Recruiting | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Collaborators: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Fabio Martelli, Dr, PhD, Molecular Cardiology Laboratory Director, IRCCS Policlinico S. Donato
Other Study IDs: RNA-HF-AS
Record Dates: First submitted 2017-07-17; First posted 2017-08-31 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure; Aortic Stenosis
Keywords: miRNA; lncRNAs; transcriptome; heart failure; aortic stenosis; biomarkers
MeSH Terms: conditions — Heart Failure; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — cardiac tissue and blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Non end-stage heart failure: Measurement of RNAs in non end-stage heart failure patients undergoing to left ventricle reconstruction
  Interventions: Diagnostic Test: measurement of RNAs
- End-stage heart failure: Measurement of RNAs in end-stage heart failure patients undergoing to left ventricular assisted device (LVAD)
  Interventions: Diagnostic Test: measurement of RNAs
- Aortic Stenosis: Measurement of RNAs in patients affected by cardiac hypertrophy leading to aortic stenosis and requiring cardiac myectomy
  Interventions: Diagnostic Test: measurement of RNAs
- Controls: Measurement of RNAs in individuals not affected by cardiovascular diseases
  Interventions: Diagnostic Test: measurement of RNAs

INTERVENTIONS:
Diagnostic Test: measurement of RNAs

SUMMARY:
This study is aimed to investigate the global transcriptome in order to determine the expression profile of messenger RNAs (mRNAs), as well as long noncoding- (lncRNAs) and micro noncoding-RNAs (miRNAs) in heart failure (HF) and in aortic stenosis (AS). The aim is to clarify their role in cardiac disease pathogenesis, as well as their potential as biomarkers. To this purpose, both tissue and blood specimens will be collected and patients will be compared to individuals not affected by cardiovascular diseases.

DETAILED DESCRIPTION:
The investigators will collect plasma and cardiac tissue specimens from consenting subjects. The investigators will evaluate the expression of mRNAs, miRNAs and lncRNAs in patients affected by both end-stage and not end-stage HF as well as in patients affected by aortic stenosis and undergoing valve replacement and requiring cardiac myectomy. The tissue dysregulated RNAs will be next measured in plasma samples in order to clarify their potential as biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Non end-stage heart failure

   * left ventricle restoration surgery (SVR)
   * End Systolic Volume Index (ESVI) >35 ml/m2
   * Ejection Fraction (EF)<40%
   * previous transmural anterior myocardial infarction (MI)
   * age: 40-75
2. End-stage heart failure

   * left ventricle assisted device (LVAD) surgery
   * age: 40-75
   * Ejection Fraction (EF) <25%
   * End Systolic Volume Index (ESVI)≥60 ml/m2
3. Aortic Stenosis

   * aortic valve replacement
   * intracardial pressure difference >40 mmHg
   * septal diameter ≥1.3 cm

Exclusion Criteria:

1. Non end-stage heart failure

   * End Systolic Volume Index (ESVI)<35 ml/m2
   * Ejection Fraction (EF)>40%
   * Time from MI unknown
   * Pregnancy
   * Other genetic diseases
   * Neoplasms
   * Collagenopathies
   * Chemo/radiotherapy
   * Prolonged use of corticosteroids
   * Infections
   * Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV) (not vaccination) and Hepatitis C Virus (HCV) positive
2. End-stage heart failure

   * EF>25%
   * Time from MI unknown
   * Pregnancy
   * Other genetic diseases
   * Neoplasms
   * Collagenopathies
   * Chemo/radiotherapy
   * Prolonged use of corticosteroids
   * Infections
   * Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV) (not vaccination) and Hepatitis C Virus (HCV) positive
3. Aortic Stenosis

   * coronaropathies
   * Pregnancy
   * Other genetic diseases
   * Neoplasms
   * Collagenopathies
   * Chemo/radiotherapy
   * Prolonged use of corticosteroids
   * Infections
   * Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV) (not vaccination) and Hepatitis C Virus (HCV) positive

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac surgery patients
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-05-30 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac tissutal mRNAs signatures | from Year 1 to Year 3
  The mRNAs cardiac tissutal signatures of non- and end-stage heart failure patients and of aortic stenosis patients compared to controls
Cardiac tissutal miRNAs signatures | from Year 1 to Year 3
  The miRNAs cardiac tissutal signatures of non- and end-stage heart failure patients and of aortic stenosis patients compared to controls
Cardiac tissutal lncRNAs signatures | from Year 1 to Year 3
  The lncRNAs cardiac tissutal signatures of non- and end-stage heart failure patients and of aortic stenosis patients compared to controls

SECONDARY OUTCOMES:
Non end-stage, end-stage heart failure, aortic stenosis mRNAs signatures in plasmas | from Year 3 to Year 5
  The mRNAs dysregulated in cardiac tissues will be measured in blood plasma samples of non- and end-stage heart failure patients and of aortic stenosis patients compared to controls
Non end-stage, end-stage heart failure, aortic stenosis miRNAs signatures in plasmas | from Year 3 to Year 5
  The miRNAs dysregulated in cardiac tissues will be measured in blood plasma samples of non- and end-stage heart failure patients and of aortic stenosis patients compared to controls
Non end-stage, end-stage heart failure, aortic stenosis lncRNAs signatures in plasmas | from Year 3 to Year 5
  The lncRNAs dysregulated in cardiac tissues will be measured in blood plasma samples of non- and end-stage heart failure patients and of aortic stenosis patients compared to controls

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Martelli, Dr, Principal Investigator — IRCCS Policlinico S. Donato
Locations (2):
- Italy (2):
  - Irccs Policlinico San Donato, San Donato Milanese, Milan
  - Ospedale San Raffaele, Milan

IPD SHARING:
Plan to Share IPD: No